CLINICAL TRIAL: NCT04605458
Title: Contingency Management to Promote Smoking Abstinence in Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00099446; R01CA251158-01 (NIH)
Record Dates: First submitted 2020-09-25; First posted 2020-10-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contingency Management (Experimental)
  Interventions: Combination Product: Contingency Management
- Standard Care (Active Comparator)
  Interventions: Combination Product: Standard Care

INTERVENTIONS:
Combination Product: Contingency Management — Participants will receive 3-6 counseling sessions, nicotine patches & lozenges, and monetary payment delivered contingent on abstinence verified by CO breath test.
  Arms: Contingency Management
Combination Product: Standard Care — Participants will receive 3-6 counseling sessions, nicotine patches & lozenges, and CO breath test monitoring.
  Arms: Standard Care

SUMMARY:
This is a smoking cessation treatment study. Patients who have a cancer or a suspected cancer who will undergo surgical removal of their cancer are eligible to participate in this study. A novel smoking cessation treatment will be provided to half of the participants in the study. All study participants will receive standard smoking cessation therapy including counseling and the nicotine patch.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. smoking 1 or more combustible tobacco products per day
3. diagnosed with or suspicion of any type of operable cancer

Exclusion Criteria:

1. unstable psychiatric/medical conditions such as suicidal ideation, acute psychosis, or dementia
2. non-English speaking
3. use of alternative nicotine delivery systems (e.g., e-cigarettes, snus, etc)
4. pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Abstinence Rates as assessed by self-report for past 7 days, Carbon Monoxide Breath Monitoring and/or Anabasine testing | Changes between the study intake appointment to day of surgery, up to five weeks apart
  Abstinence will be defined by 7 days by self-report of no tobacco products, confirmed by CO breath test less than or equal to 4ppm and/or urine anabasine levels less than or equal to 2 ng/ml

SECONDARY OUTCOMES:
Abstinence Rates as assessed by self-report for past 7 days, Carbon Monoxide Breath Monitoring and/or Anabasine testing | Three and Six months after surgery date
  Abstinence will be defined by 7 days by self-report of no tobacco products, confirmed by CO breath test less than or equal to 4ppm and/or urine anabasine levels less than or equal to 2 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rojewski AM, Fucito LM, Baker NL, Palmer AM, Foster MG, Warren GW, Bernstein SL, Toll BA. Preoperative contingency management intervention for smoking abstinence in cancer patients: trial protocol for a multisite randomised controlled trial. BMJ Open. 2021 Jun 29;11(6):e051226. doi: 10.1136/bmjopen-2021-051226. PMID 34187835

DOCUMENTS (1):
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04605458/ICF_001.pdf